CLINICAL TRIAL: NCT00317343
Title: RIAPRE - A Non-interventional Registry on the Anticoagulation Treatment in High Risk Elective Percutaneous Coronary Interventions
Brief Title: RIAPRE - Non-interventional Registry of Anticoagulation Treatment (BI-006-IT)
Status: Withdrawn | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Nycomed
Other Study IDs: BI-006-IT
Record Dates: First submitted 2006-03-30; First posted 2006-04-24 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Disease
Keywords: Patients candidate to a PCI with a planned anticoagulation regime other than unfractionated heparin in monotherapy
MeSH Terms: conditions — Coronary Disease | interventions — bivalirudin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bivalirudin (thrombin specific anticoagulant) — Percutaneous Coronary Intervention

SUMMARY:
RIAPRE is a non-interventional registry to be settled in Italy with the purpose of collecting data on 600 cases of high risk elective percutaneous coronary intervention (PCI) patients treated with an anticoagulation regime different from unfractionated heparin in monotherapy. About thirty catheterization laboratories will co-operate in this activity. The long term outcome of patients will be taken into consideration. The availability of these data will allow for a better understanding of the therapeutic needs in this area.

ELIGIBILITY:
Inclusion Criteria :

* Medical condition or disease to be studied: age > 18 years.
* Patients are candidates for a PCI with a planned anticoagulation regime other than unfractionated heparin in monotherapy. Taking into consideration the national and international guidelines for this area and the registered indications of the drugs currently used for this purpose it is predicted that the patients will probably receive one of the following:

  * unfractionated heparin as an intravenous (IV) bolus followed by IV bolus + infusion of a GPI (abciximab, tirofiban or eptifibatide); or
  * bivalirudin as an IV bolus followed by IV infusion, as per the pertinent Summary of Product Characteristics (SPCs).
* Having provided an informed consent (to anonymous data treatment).
* A planned anticoagulation regime means that any candidate patient should be identified on the basis of pre-procedural factors and requested to give his/her consent before the PCI is initiated. Patients receiving bail-out GPI for intraprocedural complications should NOT be considered for the inclusion. However, a pre-included patient could receive a bail-out GPI if deemed necessary.
* The allocation of any individual patient to the category of "high risk" elective PCI will be made independently and autonomously by the caring physician. However, it is recommended to consider the suitability of patients on the basis of these indicative elements:

  * age > 75 years.
  * known diabetes mellitus (type I or type II).
  * known renal insufficiency, i.e. serum creatinine > 1.8 mg or glomerular filtration rate (GFR) > 60 ml/min (calculated with the Cockroft formula).
  * multivessel or complex procedure.
  * planned stent on a bifurcation.
  * planned stent > 6 cm long.
  * PCI on a degenerated venous bypass: in this particular case a distal protection device should always be used.
  * non ST elevation acute coronary syndrome with a PCI planned later than 72 hours after the diagnosis without clinical instability (= "cooled" non ST elevation acute coronary syndrome). This type of patient is considered to be essentially stable and his/her level of risk can be comparable to the risk of patients who are candidates for elective PCI with additional risk factors as listed above.

Exclusion Criteria:

* There will be no specific exclusion criteria other than those listed in the Summary of Product Characteristics of every individual agent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-03; Study Completion 2008-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Project Management, Study Chair — Headquarters